CLINICAL TRIAL: NCT06721377
Title: Clinical and Radiographic Evaluation of Different Attachments on Implant-Retained Mandibular Overdenture.
Brief Title: Evaluation of Different Attachments on Implant-Retained Mandibular Overdenture.
Acronym: Overdenture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Sara Hossam El-din Kadry Othman, Assistant lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC al azhar university
Record Dates: First submitted 2024-11-30; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Edentulism in Lower Jaw; Edentulism
Keywords: overdenture; implant placemnent; Novaloc attachment.; Equator attachment; edentulism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (Active Comparator): Equator attachment
  Interventions: Procedure: Novaloc attachment
- study (Experimental): Novaloc attachment
  Interventions: Procedure: Equator attachment

INTERVENTIONS:
Procedure: Novaloc attachment — upper complete dentures and lower complete overdentures. The upper complete denture will be mucosa supported and the lower complete denture will be supported and retained for all patients by two dental implants in the inter-foraminal region & will be loaded by Novaloc attachment.
  Arms: control
Procedure: Equator attachment — upper complete dentures and lower complete overdentures. The upper complete denture will be mucosa supported and the lower complete denture will be supported and retained for all patients by two dental implants in the inter-foraminal region& will be loaded by Equator attachment.
  Arms: study

SUMMARY:
Patients will be selected from the outpatient clinic of Removable Prosthodontic Department. Faculty of Dental Medicine for Girls, Al-Azhar University..

Each patient will be assessed for eligibility and Informed consent will be obtained from patient after explanation of the treatment protocols and expected outcomes or alternative management.

DETAILED DESCRIPTION:
All 10 patients will receive upper complete dentures and lower complete overdentures. The upper complete denture will be mucosa supported and the lower complete denture will be supported and retained for all patients by two dental implants in the inter-foraminal region. Patients will be divided into two groups, one group will be loaded by Novaloc attachment. While the other group will be loaded by Equator attachment. Implants will be functionally loaded after three months of insertion.

ELIGIBILITY:
Inclusion Criteria:

* All patients' ridges should be covered with firm mucosa which is free from any signs of inflammation or ulceration.
* Patients should be free from any bone disorder and exhibit adequate height and width of the residual alveolar ridge.
* All patients must have sufficient inter arch space.

Exclusion Criteria:

* Patients with oral or systemic diseases.
* Patients with xerostomia or excessive salivation.
* Patients with parafunctional habits (bruxism or clenching).
* Heavy smoker or alcoholic patients.
* Patients with history of temporo-mandibular dysfunction.
* Patients with brain disorders or psychiatric disorders.

Ages: 65 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic evaluation of bone height | at baseline, 6 and 12 months
  Radiographic evaluation of bone height around each implant and at distal extension area will be evaluated using cone beam CT (CBCT)
Radiographic evaluation of bone density | at baseline, 6 and 12 months
  Radiographic evaluation of bone density around implant and at distal extension area will be evaluated using cone beam CT (CBCT)

SECONDARY OUTCOMES:
Pocket depth | at baseline, 6 and 12 months
  Pocket depth will be measured using periodontal probe

CONTACTS AND LOCATIONS:
Overall Officials: sara H kadry, masters, Principal Investigator
Locations (1):
- Faculty of Dental Medicine , Al Azhar Univeristy For Girls, Cairo, Nasr City - Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No